CLINICAL TRIAL: NCT04425122
Title: The Microbiome of Oesophageal Squamous Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Hon Chi Yip, Associate Consultant, Chinese University of Hong Kong
Other Study IDs: CRE-2020.186
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Esophageal Cancer; Microbial Colonization
Keywords: Esophageal squamous cell carcinoma; Microbiome
MeSH Terms: conditions — Esophageal Neoplasms; Communicable Diseases; Esophageal Squamous Cell Carcinoma | interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Oral and esophageal rinse
  2. Biopsy samples from oesophageal cancer, adjacent non-cancer mucosa, as well as random oesophageal biopsies from healthy individuals
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Esophageal cancer: Patients with esophageal cancer (SCC)
  Interventions: Diagnostic Test: Upper endoscopy
- Non-cancer group: Non-cancer patients scheduled for upper endoscopy
  Interventions: Diagnostic Test: Upper endoscopy

INTERVENTIONS:
Diagnostic Test: Upper endoscopy — Upper endoscopy would be performed. Biopsy would be taken from oesophageal cancer tissue and adjacent non-cancerous mucosa
  Groups: Esophageal cancer
Diagnostic Test: Upper endoscopy — Upper endoscopy would be performed. Random biopsy would be taken from normal non-cancer esophageal mucosa.
  Groups: Non-cancer group

SUMMARY:
This is a prospective study on the microbiota associated with oesophageal squamous cell carcinoma (SCC). Patients with newly diagnosed SCC of oesophagus would be recruited for taking samples of oral and oesophageal rinse, tissue biopsies for investigation of the microbiota of oesophageal cancer. Control patients would be identified from patients scheduled for routine endoscopy.

DETAILED DESCRIPTION:
Oesophageal carcinoma significantly contributes to the global cancer burden ranking as the sixth leading cause of global cancer-related death. Oesophageal squamous cell carcinoma (OESCC) is one of the most common type of upper gastrointestinal (UGI) carcinoma in some regions globally, particularly China and Japan in Asia. The disease has an extremely poor prognosis, with overall 5-year survival rates of less than 30%, mainly due to late stage at diagnosis and high likelihood of distant metastases. Although OESCC is associated with risk factors including smoking and alcohol, the aetiology of OESCC is still poorly understood.

Increasing evidence indicates a key role for bacterial microbiota in carcinogenesis. Emerging data implicates the human microbiome in a variety of cancers, most notably Fusobacterium in colorectal cancer and Helicobacter in gastric cancer. The consortium of bacterial microbiome colonizing the gastrointestinal tract is extensive and interact in a complex manner. The microbiome may interact with genetic and environmental factors to metabolize dietary constituents and xenobiotics, among other functions. When the microbial balance is disturbed, the microbiota could alter host cell proliferation and death, manipulate the immune system, and influence host metabolism, giving rise to carcinoma. Several studies have reported an important role of the human microbiota in upper gastrointestinal carcinoma and found associations between the microbiota and some diseases of the UGI tract, such as esophagitis and Barrett esophagus, and with squamous dysplasia and squamous carcinoma of the oesophagus. Another even less well known is the role of the fungal microbiome in OESCC.

Here the investigators will seek to evaluate the role of the bacterial and fungal microbiome in OESCC and the host microbe interactions that may play a role in the understanding and management of OESCC.

Study questions:

1. Does the microbiome differ between OESCC and normal patients?
2. Does the microbiome change from normal through premalignancy to malignancy?
3. What are the mechanisms involved in the microbiome and the development or progression of OESCC?

Study design:

This is a prospective study. The study will be carried out in accordance with the Declaration of Helsinki.

Patients would be recruited from the Prince of Wales Hospital from Jun 2020 to May 2025. 100 patients with newly diagnosed OESCC or oesophageal squamous dysplasia will be recruited to the test group. 100 patients undergoing an oesophagogastroduodenoscopy (OGD) without a history of malignancy will be recruited to the control group. The expected duration of subject participation is less than two months.

The study has two visits, as follows:

1. Visit 1:

   i. To discuss about the project and to sign the informed consent form; ii. To collect oral rinse 20ml; iii. To complete questionnaire: Gut Microbe - Medical and health questionnaire.
2. Visit 2:

To have OGD. Visit 2 will be performed within two months post Visit 1 and must before treatment.

i. Test group: With examination of the lesion with biopsy of tumor, biopsy of adjacent normal tissue, flush with normal saline.

ii. Control group: Will have a biopsy of normal tissue and flush with normal saline.

Sample size justification:

This is a prospective study with no previous data based on OESCC. But based on data from head and neck squamous cell carcinoma (HNSCC) with some overlap in traditional risk factors the investigators target to recruit at least 100 OESCC patients and 100 healthy subjects. In HNSCC study using 54 HNSCC tumour tissues and the adjacent normal tissues has generated 16S rRNA short reads able to discriminate cases from controls. A total of 77 bacterial genera with >0.1% mean relative abundance was observed in tumour tissues. A rarefaction analysis indicated that at least 73 genera can be detected from any of 35 samples, suggesting that recruitment of 100 patients and 100 controls meets the minimized sample size to contain nearly full spectrum of oral bacteria and is expected to have a power of 0.8 and confidence level of 95% to characterize oral microbiota dysbiosis between cases and controls.

Independent variables

The following independent variables will be examined to evaluate the association of the methylation panel and OESCC:

1. Clinical factors: TNM staging of disease, comorbidities;
2. Cancer risk factors: smoking history, alcohol consumption;
3. Patient factors: sex, age;
4. Histologic characteristics: tumour depth, extracapsular spread, lymphovascular invasion, perineural invasion.

Samples:

Oral rinse: Before the procedure, an oral rinse would be performed by asking all patients to rinse the oral cavity with 20ml normal saline. The resultant solution would be kept for subsequent analysis.

Endoscopic procedures Endoscopic procedures would be performed by doctors with expertise on performing upper endoscopy. It would be conducted at the Combined Endoscopy Center, Prince of Wales Hospital. Topical local anaesthetic will be applied to the oropharynx. Endoscopes with magnification /dual focus and NBI function would be used. A soft black hood would be attached to the tip of the endoscope for better focal length adjustment.

Patients in the test group would then undergo endoscopy with one biopsy of the tumor and one biopsy of the adjacent normal esophageal mucosa. In addition, oesophageal rinse would also be performed by flushing the esophagus gently with 20ml normal saline and the fluid suctioned and collected for analysis.

Patients in the control group would undergo endoscopy as per usual clinical practice. One biopsy would be taken from normal esophageal mucosa for analysis. Similarly, oesophageal rinse would be performed.

Experiments DNA extraction and bisulphite modification: DNA from microdissected fresh tissues and saliva will be extracted with phenol-chloroform, precipitated in 100% ethanol, centrifuged at 5100 rpm for 45 minutes, washed in 70% ethanol twice, dissolved in LoTE buffer (10mM TRIS hydrochloride, 1mM EDTA buffer, pH 8), and stored at -80°C.

RNA extraction: Fresh tissue will be stored in RNAlater for extraction of RNA and stored in -80°C.

Genomic analysis: Utilizing next generation sequencing analysis for copy number aberrations and single nucleotide variations to analyse the samples collected using shotgun massive parallel sequencing as previously described. We will also use sequencing to analyse the microbiota of the cohort. Bacterial 16S rRNA gene sequencing: An aliquot of DNA will be used to screen oral microbial community using 16S rRNA gene V3- V4 region amplicon sequencing 24. QIIME2 with the latest Silva ribosomal RNA database will be used to classify amplicon sequence variant, with operational taxonomic table showing the proportion of bacterial reads per sample. Mycobiota ITS gene sequencing: we will target mycobiota internal transcribed spacer gene (ITS) to characterize oral fungal community. A short region of ITS1 (~270 bp) will be PCR amplified and sequenced using MiSeq. The reads will be processed against a fungal UNITE database, and the classification tables will be generated at the species-, genera- and OTU-level for statistical analyses.

Expression analysis: The investigators will determine if these genomically altered tumors express specific changes in signaling proteins using immunohistochemical staining (IHC) and protein profiling by protein arrays. FFPE-sections or frozen tissues will be harvested for alongside with genomic characterization study for IHC analyses, or protein profiling. For IHC analysis or protein profiling, a total of 5 FFPE-slides will be employed for IHC or protein extraction for protein profiling as previously published. RNA will be extracted and subjected to RNA analyses, including RNA-seq, expression array and RT-PCR analyses so as to determine specific gene expression patterns of oesophageal tumors, as well as expression of potential biomarkers.

Bacterial Culture: To further understand the role of the microbiome as a biomarker in OESCC tissue specimens will be cultured for bacteria identified in sequencing to be significantly enriched in tumours. Tissue specimens were aseptically macerated with disposable scalpels and vortexed for 30 seconds in PBS (500 l), and the neat suspensions were used to make 10-fold 2 ) dilutions. Neat suspensions (50 l) were each spread onto blood agar (BA), fastidious anaerobe agar (FAA) (BA and FAA supplemented with 5% defibrinated sheep blood; TCS Biosciences Ltd.), and Sabouraud's agar (Lab MTM; International Diagnostics Group plc). The dilutions and final PBS washes of the specimens (see above) were spread onto BA and FAA. BA and Sabouraud's agar plates were incubated aerobically at 37°C for 48 h. FAA plates were incubated in an anaerobic cabinet at 36°C for 96 h.

Outcomes measures

1. Loco-regional recurrence free survival will be recorded from time of diagnosis to time of recurrence locally, regionally or local and regionally.
2. Disease specific survival will be recorded from time of diagnosis to time of death from OESCC.
3. Overall survival will be recorded from time of diagnosis to time of death from all causes.

Statistical Analysis Association between microbes, surgery treatment, and individuals' metadata (e.g., gender, age, smoking, drinking, T/N stages, survival, recurrence) will be analysed using a mix of ordination, non-parametric multivariate analysis of variance, matrix correlation, chi-square test, generalized linear model, or conditional logistic regression models. The performance of the final biomarkers will be assessed by cross-validation and summarized by c-index score to assess the concordance between model and comparison groups using ROC curves. All multiple testing corrections will be performed by computing FDRs using the BenjaminiHochenberg method, and adjusted p values < 0.05 will be considered statistically significant.

ELIGIBILITY:
Cancer group:

Inclusion criteria:

1. 18 Years and older
2. Able to provide informed consent
3. No cognitive impairment
4. Newly diagnosed OESCC or oesophageal dysplasia.

Exclusion Criteria:

1) On anticoagulation including Plavix, warfarin and NOAC's

Control group:

Inclusion Criteria:

1. Patients undergoing an OGD without a history of malignancy
2. 18 Years and older
3. Able to provide informed consent
4. No cognitive impairment

Exclusion Criteria:

1) On anticoagulation including Plavix, warfarin and NOAC's

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General Inclusion Criteria for both study groups, Test group and Control group.
  1. 18 Years and older
  2. Able to provide informed consent
  3. No cognitive impairment
  General Exclusion Criteria for both study groups, Test group and Control group.
  1) On anticoagulation including Plavix, warfarin and NOAC's
  Test group:
  Additional Specific Inclusion Criteria:
  1) Newly diagnosed OESCC or oesophageal dysplasia.
  Control group:
  Additional Specific Inclusion Criteria:
  1) Patients undergoing an OGD without a history of malignancy
  Withdrawal criteria:
  1. The subject withdraws consent.
  2. If the subject is non-cooperative and/ or undisciplined.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbiological culture from biopsy specimens | 1month
  Pattern of culture from specimens obtained, compared between cancer and non-cancer

SECONDARY OUTCOMES:
Loco-regional recurrence free survival | 5 year
  Time of diagnosis to time of recurrence locally, regionally or local and regionally.
Disease specific survival | 5 year
  Time of diagnosis to time of death from OESCC.
Overall survival | 5 year
  Time of diagnosis to time of death (All cause)

CONTACTS AND LOCATIONS:
Overall Officials: Hon Chi Yip, FRCSEd, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided